CLINICAL TRIAL: NCT04557865
Title: Establishing 18F PMPBB3 (APN 1607) PET Imaging, Genetic and Plasma Biomarkers for Risk Identification, Disease Progression and Prognosis of Tauopathy Related Parkinsonism s Yndromes
Brief Title: Establishing 18F PMPBB3 (APN 1607) PET Imaging Markers for Diagnosis of Tauopathy Parkinsonism Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202006181MINB
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Tau Distributions in Patients With Tauopathy Using APN-1607 PET Scan
Keywords: Tau
MeSH Terms: conditions — Pick Disease of the Brain | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receving 18F-PMPBB3 (APN-1607) PET imaging (Experimental): Single arm, open label
  Interventions: Diagnostic Test: 18F-PMPBB3 (APN-1607) PET imaging

INTERVENTIONS:
Diagnostic Test: 18F-PMPBB3 (APN-1607) PET imaging — 1. Name: 18F-PMPBB3 (APN-1607, MNI-958, or APN-0000455)
  2. Dosage form: injection form
  3. Strength: 5mCi/dose
  4. Dosage and administration: 5mCi, intravenous injection
  5. Mechanism of action (if known): bind to tau protein in the brain
  6. Pharmacological category: radiopharamceutical

SUMMARY:
Parkinson's disease (PD) is one of the most common neurodegenerative disorders. The diagnosis of PD is primarily based on clinical presentations while the pathology stage of a-synuclein containing Lewy body deposition has already advanced. In addition to PD, there is another group of patients presenting with parkinsonism features mixed with other neurodegenerative symptoms. Pathologically, patients with these PD-mimicking parkinsonism syndromes, such as progressive supranuclear palsy (PSP), corticobasal degeneration disorders (CBGD) and frontotemporal dementia (FTD) with/without parkinsonism, have 4 repeat paired helical filament forms of tau protein (4R PHF-tau) aggregations in the neurons. Patients with these tauopathy related parkinsonism-plus syndromes could initially present as PD symptoms but will have a more deliberating disease course and combine with other systems degeneration. These patients are often a substantial diagnostic challenge to clinicians. Therefore, there is an urgent need to develop reliable imaging and biofluid biomarkers for differentiating patients with PD and variable parkinsonism-plus syndromes.

Recently, new generation of novel radiotracer 18F-PMPBB3 (APN-1607), which can be labeled with 4R PHF-tau without significant off-target binding, has been successfully developed. Therefore, this study will enroll 150 participants, including 30 healthy controls, 30 PD patients, and 60 patients with different parkinsonism-plus syndromes (including 10 patients with multiple system atrophy, 10 patients with progressive supranuclear palsy, 10 patients with cortical basal syndrome and 30 patients with frontotemporal dementia), and 30 patients with mild cognitive decline (MCI) or Alzheimer's disease (AD). All participants will receive complete neurological examination, 18F-PMPBB3 (APN-1607) PET, brain MRI scans, plasma markers for total/phosphorylated tau, a-synuclein and Ab42/Ab40 and genetic markers covering MAPT、SNCA、LRRK2、GBA and APOE genes. We aim to explore:

1. Whether 18F-PMPBB3 (APN-1607) can differentiate patients with tauopathy (PSP, CBGD, FTD, MCI and AD) and synucleinopathy (PD, MSA).
2. Whether the distribution of tau deposition detected by 18F-PMPBB3 (APN-1607) correlate to disease severity, progression, and prognosis in patients with tauopathy.
3. Whether the loading of tau deposition detected by 18F-PMPBB3 (APN-1607) correlate to plasma levels of total/phosphorylated tau.
4. Determine specific genetic susceptibility sub-groups are more vulnerable to tau deposition detected by 18F-PMPBB3 (APN-1607) in patients with tauopathy.

The research results will help to understand the potential of 18F-PMPBB3 (APN-1607) as an imaging biomarker for diagnosis, severity and therapeutic assessment tool for patients with tauopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Patients fulfill the criteria of United Kingdom Brain Bank Diagnostic Criteria of "possible" or "probably" PD.
3. Patients fulfill the criteria of MDS consensus criteria of "possible" or "probably" MSA.
4. Patients fulfill the criteria of NINDS-SPSP clinical criteria for the diagnosis of PSP "as possible" or "probably" PSP, and healthy volunteer with no clinically relevant finding on physical examination at screening visit.
5. Patients fulfill the criteria of Work Group on Frontotempotal Dementia and Pick's Disease of "possible" or "probably" FTD.
6. Patients fulfill the Armstrong's criteria of "possible" or "probably" CBGD.
7. Patients fulfill the National Institute on Aging-Alzheimer's Association (NIA-AA) workgroup for clinical diagnostic guidelines (NIA-AA-C) for MCI.
8. Patients fulfill the National Institute on Aging-Alzheimer's Association (NIA-AA) workgroup for clinical diagnostic guidelines (NIA-AA-C) for AD.
9. Neurologically normal controls.
10. Age range 20-90 years

Exclusion Criteria:

1. Implantation of metal devices including cardiac pacemaker, intravascular metal devices.
2. Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes, acute myocardial infarction, poorly controlled diabetes, previous head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases
3. Major psychiatric disorders, drug or alcohol abuse and major depression
4. Pregnant women or breast- feeding women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
The distribution of tau measured by Standardized Uptake Value Ratio (SUVR) as Assessed by 18F-PM-PBB3 tau PET Scan | 1.5 years
  Tau Distribution among patients with parkinsonism-plus syndromes, Parkinson's disease (PD), Alzheimer's disease (AD) spectrum, and normal controls measured by Standardized Uptake Value Ratio (SUVR) as Assessed by 18F-PM-PBB3 tau PET Scan

SECONDARY OUTCOMES:
The amount of tau measured by SUVR as assessed by 18F-PM-PBB3 tau PET Scan as disease severity in patients with tauopathy parkinsonism-plus syndrome | 1.5 years
  The correlation between Tau distribution among patients with tauopathy parkinsonism-plus syndrome with clinical severity.
The amount of tau measured by SUVR as assessed by 18F-PM-PBB3 tau PET Scan as disease progression in patients with tauopathy parkinsonism-plus syndrome. | 1.5 years
  The correlation between Tau distribution among patients with tauopathy parkinsonism-plus syndrome with clinical progression speed.
To correlate the loading of tau deposition detected by 18F-PMPBB3 (APN-1607) correlate to plasma levels of total/phosphorylated tau. | 1.5 years
  The correlation between Tau distribution among patients with tauopathy parkinsonism-plus syndrome with plasma levels of total/phosphorylated tau.
To determine specific genetic susceptibility sub-groups are more vulnerable to tau deposition detected by 18F-PMPBB3 (APN-1607) in patients with tauopathy. | 1.5 years
  The correlation between Tau distribution among patients with tauopathy parkinsonism-plus syndrome with genetic variants of candidate genes.
Safety endpoints - ECG | 1.5 years
  Changes of electrocardiography (ECG) QT Interval before and after receiving 18F-PMPBB3 (APN-1607) scans.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1.5 years
  Any discomfort after receiving 18F-PMPBB3 (APN-1607) scans.
Safety endpoints-Vital signs | 1.5 years
  Changes of blood pressure (changes of SBP >=20 mmHg) before and after receiving 18F-PMPBB3 (APN-1607) scans.
Safety endpoints-adverse event assessments | 1.5 years
  Any discomfort after receiving 18F-PMPBB3 (APN-1607) scans.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hsien Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No